CLINICAL TRIAL: NCT00427570
Title: A Clinical Trial to Evaluate Postoperative Immunotherapy and Postoperative Systemic Chemotherapy in the Management of Resectable Colon Cancer
Brief Title: Fluorouracil, Semustine, and Vincristine Compared With BCG in Treating Patients With Dukes' B or Dukes' C Colon Cancer That Has Been Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000071312; NSABP-C-01
Record Dates: First submitted 2007-01-18; First posted 2007-01-29 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2010-08

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — BCG Vaccine; Biological Therapy; Fluorouracil; Semustine; Vincristine

INTERVENTIONS:
Biological: BCG vaccine
Biological: biological therapy
Drug: fluorouracil
Drug: semustine
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vincristine, fluorouracil, and semustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapies, such as BCG, may stimulate the immune system in different ways and stop tumor cells from growing. It is not yet known whether combination chemotherapy is more effective than BCG in treating colon cancer that has been removed by surgery.

PURPOSE: This randomized phase III clinical trial is studying giving fluorouracil together with semustine and vincristine to see how well they work compared with giving BCG in treating patients with Dukes' B or Dukes' C colon cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Obtain information to define subsets of colon cancer patients at high risk of recurrence. II. Correlate pathologic and biologic parameters with disease-free interval and survival. III. Determine the value of surgical and ancillary techniques in management of colon cancer. IV. Compare disease-free interval and survival after curative resection vs. chemotherapy with 5-fluorouracil/methyl-CCNU/vincristine vs. BCG immunotherapy. V. Relate the total lymphocyte count to the course of the disease. VI. Determine the feasibility of conducting a trial employing immunotherapy in a surgical adjuvant setting. VII. Identify appropriate future protocols based on data generated in the study.

OUTLINE: Randomized study for patients with Dukes Stage B and C disease only. All patients with Dukes A and D lesions enter Arm I. Arm I: No therapy following surgery. Arm II: 3-Drug Combination Chemotherapy. 5-Fluorouracil, 5-FU, NSC-19893; Methyl-CCNU, MeCCNU, NSC-95441; Vincristine, VCR, NSC-67574. Arm III: Immunotherapy. BCG-Pasteur, BCG, NSC-B116328.

PROJECTED ACCRUAL: Protocol closed February 1984.

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: See General Eligibility Criteria

Max Age: 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1977-09; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Study Chair — Allegheny Cancer Center at Allegheny General Hospital

REFERENCES:
- [Background] O'Connell MJ, Lavery I, Yothers G, Paik S, Clark-Langone KM, Lopatin M, Watson D, Baehner FL, Shak S, Baker J, Cowens JW, Wolmark N. Relationship between tumor gene expression and recurrence in four independent studies of patients with stage II/III colon cancer treated with surgery alone or surgery plus adjuvant fluorouracil plus leucovorin. J Clin Oncol. 2010 Sep 1;28(25):3937-44. doi: 10.1200/JCO.2010.28.9538. Epub 2010 Aug 2. PMID 20679606
- [Background] Wilkinson NW, Yothers G, Lopa S, Costantino JP, Petrelli NJ, Wolmark N. Long-term survival results of surgery alone versus surgery plus 5-fluorouracil and leucovorin for stage II and stage III colon cancer: pooled analysis of NSABP C-01 through C-05. A baseline from which to compare modern adjuvant trials. Ann Surg Oncol. 2010 Apr;17(4):959-66. doi: 10.1245/s10434-009-0881-y. PMID 20082144
- [Background] Wilkinson NW, Yothers G, Lopa SH, et al.: Long-term survival results of surgery alone compared with surgery plus 5-fluorouracil and leucovorin for stage II and stage III colon cancer: pooled analysis of NSABP adjuvant trials C-01 through C-05. [Abstract] American Society of Clinical Oncology 2009 Gastrointestinal Cancers Symposium, 15-17 January 2009, San Francisco, CA. A-442, 2009.
- [Background] Kim GP, Colangelo LH, Wieand HS, Paik S, Kirsch IR, Wolmark N, Allegra CJ; National Cancer Institute. Prognostic and predictive roles of high-degree microsatellite instability in colon cancer: a National Cancer Institute-National Surgical Adjuvant Breast and Bowel Project Collaborative Study. J Clin Oncol. 2007 Mar 1;25(7):767-72. doi: 10.1200/JCO.2006.05.8172. Epub 2007 Jan 16. PMID 17228023
- [Background] Allegra CJ, Paik S, Colangelo LH, Parr AL, Kirsch I, Kim G, Klein P, Johnston PG, Wolmark N, Wieand HS. Prognostic value of thymidylate synthase, Ki-67, and p53 in patients with Dukes' B and C colon cancer: a National Cancer Institute-National Surgical Adjuvant Breast and Bowel Project collaborative study. J Clin Oncol. 2003 Jan 15;21(2):241-50. doi: 10.1200/JCO.2003.05.044. PMID 12525515
- [Background] Fisher ER, Colangelo L, Wieand S, Fisher B, Wolmark N. Lack of influence of cytokeratin-positive mini micrometastases in "Negative Node" patients with colorectal cancer: findings from the national surgical adjuvant breast and bowel projects protocols R-01 and C-01. Dis Colon Rectum. 2003 Aug;46(8):1021-5; discussion 1025-6. doi: 10.1007/s10350-004-7275-9. PMID 12907892
- [Background] Wolmark N, Colangelo L, Wieand S. National Surgical Adjuvant Breast and Bowel Project trials in colon cancer. Semin Oncol. 2001 Feb;28(1 Suppl 1):9-13. doi: 10.1016/s0093-7754(01)90245-3. PMID 11273592
- [Background] Dignam JJ, Colangelo L, Tian W, Jones J, Smith R, Wickerham DL, Wolmark N. Outcomes among African-Americans and Caucasians in colon cancer adjuvant therapy trials: findings from the National Surgical Adjuvant Breast and Bowel Project. J Natl Cancer Inst. 1999 Nov 17;91(22):1933-40. doi: 10.1093/jnci/91.22.1933. PMID 10564677
- [Background] Mamounas E, Wieand S, Wolmark N, Bear HD, Atkins JN, Song K, Jones J, Rockette H. Comparative efficacy of adjuvant chemotherapy in patients with Dukes' B versus Dukes' C colon cancer: results from four National Surgical Adjuvant Breast and Bowel Project adjuvant studies (C-01, C-02, C-03, and C-04). J Clin Oncol. 1999 May;17(5):1349-55. doi: 10.1200/JCO.1999.17.5.1349. PMID 10334518
- [Background] Wolmark N, Fisher B, Wieand HS, Henry RS, Lerner H, Legault-Poisson S, Deckers PJ, Dimitrov N, Gordon PH, Jochimsen P, et al. The prognostic significance of preoperative carcinoembryonic antigen levels in colorectal cancer. Results from NSABP (National Surgical Adjuvant Breast and Bowel Project) clinical trials. Ann Surg. 1984 Apr;199(4):375-82. doi: 10.1097/00000658-198404000-00001. PMID 6370155
- [Background] Wolmark N, Fisher ER, Wieand HS, Fisher B. The relationship of depth of penetration and tumor size to the number of positive nodes in Dukes C colorectal cancer. Cancer. 1984 Jun 15;53(12):2707-12. doi: 10.1002/1097-0142(19840615)53:123.0.co;2-r. PMID 6722730
- [Background] Wolmark N, Cruz I, Redmond CK, Fisher B, Fisher ER. Tumor size and regional lymph node metastasis in colorectal cancer. A preliminary analysis from the NSABP clinical trials. Cancer. 1983 Apr 1;51(7):1315-22. doi: 10.1002/1097-0142(19830401)51:73.0.co;2-0. PMID 6337699
- [Background] Wolmark N, Wieand HS, Rockette HE, Fisher B, Glass A, Lawrence W, Lerner H, Cruz AB, Volk H, Shibata H, et al. The prognostic significance of tumor location and bowel obstruction in Dukes B and C colorectal cancer. Findings from the NSABP clinical trials. Ann Surg. 1983 Dec;198(6):743-52. doi: 10.1097/00000658-198312000-00013. PMID 6357118
- [Result] Smith RE, Colangelo L, Wieand HS, Begovic M, Wolmark N. Randomized trial of adjuvant therapy in colon carcinoma: 10-year results of NSABP protocol C-01. J Natl Cancer Inst. 2004 Aug 4;96(15):1128-32. doi: 10.1093/jnci/djh220. PMID 15292384
- [Result] Wolmark N, Fisher B, Rockette H, Redmond C, Wickerham DL, Fisher ER, Jones J, Glass A, Lerner H, Lawrence W, et al. Postoperative adjuvant chemotherapy or BCG for colon cancer: results from NSABP protocol C-01. J Natl Cancer Inst. 1988 Mar 2;80(1):30-6. doi: 10.1093/jnci/80.1.30. PMID 3276901
- [Result] Wolmark N, Fisher B, Rockette H, et al.: Adjuvant therapy in carcinoma of the colon: five year results of NSABP protocol C-01. [Abstract] Proceedings of the American Society of Clinical Oncology 6: A-358, 92, 1987.
- [Result] Weese JL, Starling JR, Ottery FD, et al.: Should omentectomy be part of colectomy for colon cancer? [Abstract] Proceedings of the American Society of Clinical Oncology 4: C-358, 92, 1985.